CLINICAL TRIAL: NCT04256889
Title: Use of Nfant(R) Technology Feeding System As An Adjunct To Visual Assessment And Cue-Based Feedings For Infants Born Less Than 30 Weeks Gestational Age (GA)
Brief Title: Use Of Nfant(R) Technology Feeding System For Infants Less Than 30 Weeks GA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: NFANT Labs (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RP-19-013
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Prematurity; Extreme Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Prospective case matched controlled study (not a cohort). Enrolled infants will be matched with infants in the National Medical Index based on gestational age, gender, weight and comorbidities. A two cohort, mixed regression model would be used to correlate nfant® metrics to clinical outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- nfant(R) feeding system (Experimental): Addition of nfant(R) technology, along with visual assessments and cue-based feeding practices, to facilitate an infant's progression to full oral feeding and potentially improve developmentally supportive feeding practices.
  Interventions: Device: nfant(R) feeding system

INTERVENTIONS:
Device: nfant(R) feeding system — Use of nfant(R) technology feeding system as an adjunct to visual assessment and cue-based feedings for infants born less than 30 weeks GA

SUMMARY:
The purpose of the study is to utilize the objective data provided by the nfant® suite of products, along with current NICU visual assessment and cue-based feeding practices, in order to determine if feeding performance outcomes and clinical decision making for individualized feeding plans for premature infants born less than 30 weeks PMA are impacted.

DETAILED DESCRIPTION:
Will obtain 5 official readings using the nfant(R) technology: baseline between 31 0/7 weeks and 32 0/7 weeks Post-Menstrual Age (PMA) with No Flow nipple, Cue-Based Feeding Readiness Reading with No Flow nipple no sooner than 33 0/7 weeks PMA, Post-Sequencing Reading with Extra Slow Flow nipple, Slow Flow nipple Reading, and Standard nipple Reading. The technology will also be utilized between readings 2 to 3 times a week. Phone Follow-up 2 question survey will be administered 21 days after discharge from Neonatal Intensive Care Unit.This survey entails routine questions regarding re-admission, to clarify if readmission was within 21 days of discharge, and if the reason for re-admission was feeding related.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than or equal to 29 6/7 weeks gestation at birth

Exclusion Criteria:

* Infants 30 weeks or greater gestation at birth
* Infants with known or suspected congenital anomalies or chromosomal abnormalities
* Infants with diagnoses known to interfere with oral feeding, including, but not limited to cleft lip. cleft palate, gastroschisis, Tracheoesophageal fistula, micrognathia.
* History of Intraventricular hemorrhage Grade 3 or 4 or Periventricular Leukomalacia
* Infants with known diagnoses known to interfere with Gastrointestinal absorption, including, but not limited to, Necrotizing Enterocolitis requiring surgical intervention

Ages: 22 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with decreased Feeding Related Length of Stay | up to 48 hours
  Starts when an infant can take 5 ml of breast milk or formula orally with autonomic stability
Number of participants with Full oral feeding | 33 weeks through study completion, an average of 1 year
  Gestational age at which the infant first completes 90% of minimal ordered volumes without requiring gavage feeds for a 24 hour period
Number of participants with hospital readmission for feeding related issues | Within the first 21 days after Neonatal Intensive Care Unit discharge
  Phone Follow-up
Number of inpatient Modified Barium Swallow Study (MBSS)/repeat MBSS | Neonatal Intensive Care Unit admit through study completion, an average of 1 year
  Swallow Studies
Number of participants with increased Sucking Efficiency | 31 weeks GA through study completion, an average of 1 year
  nfant(R) feeding metrics
Number of participants with increased Sucking Amplitude | 31 weeks GA through study completion, an average of 1 year
  nfant(R) feeding metrics
Number of participants with increased Sucking Frequency | 31 weeks GA through study completion, an average of 1 year
  nfant(R) feeding metrics
Number of participants with increased Sucking Duration | 31 weeks GA through study completion, an average of 1 year
  nfant(R) feeding metrics
Number of participants with increased Sucking Smoothness | 31 weeks GA through study completion, an average of 1 year
  nfant(R) feeding metrics

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Gremillion, PT, MS, CNT, Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT04256889/ICF_000.pdf